CLINICAL TRIAL: NCT06838000
Title: A Phase 3, Randomized, Modified Double-blind, Active-controlled, Parallel-group Study to Investigate the Safety and Immunogenicity of Catch-up Vaccination Regimens of a 21-valent Pneumococcal Conjugate Vaccine in Healthy Infants, Toddlers, Children, and Adolescents
Brief Title: Study of the Safety and Immunogenicity of Catch-up Vaccination With a 21-valent Pneumococcal Conjugate Vaccine (PCV21) in Healthy Infants, Toddlers, Children, and Adolescents
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSK00010; U1111-1294-7860 (Other: World Health Organization Universal Trial Number); 2024-512271-13 (Other: CTIS)
Record Dates: First submitted 2024-10-10; First posted 2025-02-20 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal Vaccines; Pneumococcal Conjugate Vaccine; Healthy Participants
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Control-Method: Active Controlled
Who Masked: Participant
Masking Description: Modified double-blind:
  * Blinding for vaccine group assignment: participants and participant's parent(s) / legally acceptable representative(s) (LARs), outcome assessors, Investigators, laboratory personnel, and Sponsor study staff
  * No blinding for vaccine group assignment: those preparing and administering the study interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Infants (7 to 11 MoA) (Experimental): Participants will receive 3 intramuscular injections of pneumococcal vaccine with an interval of:
  * 4 to 8 weeks (28 to 56 days) between the 1st dose and the 2nd dose
  * 8 to 12 weeks (56 to 84 days) between the 2nd dose and the 3rd dose AND age ≥ 12 MoA at 3rd dose
  Interventions: Biological: PCV21; Biological: 20vPCV
- Toddlers (12 to 23 MoA) (Experimental): Participants will receive 2 intramuscular injections of the pneumococcal vaccine with an interval of 8 to 12 weeks (56 to 84 days) between doses
  Interventions: Biological: PCV21; Biological: 20vPCV
- Children/adolescent (2 to 5 and 6 to 17 YoA) (Experimental): Participants will receive 1 intramuscular injection of the pneumococcal vaccine
  Interventions: Biological: PCV21; Biological: 20vPCV

INTERVENTIONS:
Biological: PCV21 — Investigational pneumococcal conjugate vaccine
Biological: 20vPCV — 20-valent pneumococcal conjugate vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of PCV21 versus 20vPCV ( 20-valent pneumococcal conjugate vaccine, Prevnar 20) for catch-up vaccination in infants (7 to 11 MoA-Months of age), toddlers (12 to 23 MoA), and children/adolescents (2 to 5 YoA and 6 to 17 YoA-years of age).

DETAILED DESCRIPTION:
The duration of each participation will be approximately 9 to 11 months for each infant participant, 8 to 9 months for each toddler participant, and 6 months for each child/adolescent participant.

ELIGIBILITY:
Inclusion Criteria:

AGE

* Aged 7 months to 17 years on the day of inclusion

TYPE OF PARTICIPANT AND DISEASE CHARACTERISTICS

* Participants who are healthy as determined by medical evaluation including medical history and physical examination

For infants (7 to 11 MoA) and toddlers (12 to 23 MoA) only

* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg or born after a gestation period above 28 (> 28 weeks) through 36 weeks with a birth weight ≥ 1.5 kg, and in both cases medically stable as assessed by the investigator

SEX, CONTRACEPTIVE/BARRIER METHOD AND PREGNANCY TESTING REQUIREMENTS For adolescents (6 to 17 YoA) only

* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:
* Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be pre-menarche or surgically sterile. OR
* Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to the study vaccine administration until at least 4 weeks after the study vaccine administration. A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 25 hours of before the first dose of study vaccine.

INFORMED CONSENT

* Assent form has been signed and dated by the participant (based on local regulations), and if applicable, and informed consent form has been signed and dated by the parent(s) or another legally acceptable representative (LAR) and by an independent witness, if required by local regulations

OTHER INCLUSIONS

* Participant and parent(s) / LAR(s) are able to attend all scheduled visits and to comply with all study procedures

Exclusion Criteria:

MEDICAL CONDITIONS

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy
* History of microbiologically confirmed S. pneumoniae infection or disease
* History of seizure or significant stable or progressive neurological disorders such as inflammatory nervous system diseases, encephalopathy, and cerebral palsy
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a product containing any of the same substances
* Laboratory-confirmed thrombocytopenia, or known thrombocytopenia, as reported by the parent(s) / LAR(s), contraindicating intramuscular (IM) injection
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of vaccine administration.

For infants (7 to 11 MoA) and toddlers (12 to 23 MoA) only

* Previous vaccination against S. pneumonia

For children (2 to 5 YoA) and adolescents (6 to 17 YoA) only

* Previous vaccination with pneumococcal polysaccharide vaccine

For adolescents (6 to 17 YoA) only

* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion

PRIOR/CONCOMITANT THERAPY

* Receipt of any vaccine in the 4 weeks preceding the vaccine administration or planned receipt of any vaccine in the 4 weeks following the vaccine administration, except for US licensed influenza vaccination, which may be received at least 2 weeks before or 2 weeks after any study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines, as applicable per local recommendations
* Receipt of immune globulins, blood or blood-derived products in the past 3 months

For children (2 to 5 YoA) and adolescents (6 to 17 YoA) only

* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw

PRIOR/CONCURRENT CLINICAL STUDY EXPERIENCE

* Participation at the time of study enrollment (or in the 6 weeks preceding the first vaccine administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure

OTHER EXCLUSIONS For adolescents (6 to 17 YoA) only

* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 7 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1268 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting immediate adverse events (AEs) | Within 30 minutes post-vaccination
  Unsolicited (spontaneously reported) systemic AEs after each and any injection of a pneumococcal vaccine
Number of participants reporting solicited injection site and solicited systemic reactions | Up to Day 7 post-vaccination
Number of participants reporting unsolicited (spontaneously reported) injection site reactions and unsolicited systemic AEs after each and any injection of a pneumococcal vaccine | Within 30 days after vaccination
Number of participants reporting serious adverse events (SAEs) and adverse events of special interest (AESIs) | From day 0 to day 517
  SAEs and AESIs are collected throughout the study period
Number of Infants (7-11 months of age [MoA]) and toddlers (12-23 MoA): with serotype-specific IgG concentrations for all serotypes included in PCV21 | On day 30 after last vaccination
  Ab (antibody) concentrations for each pneumococcal serotype are measured.
Number of Children (2-5 years of age [YoA]):with serotype specific OPA titers for all serotypes included in PCV21 | On day 30
  Serotype specific OPA titers for each pneumococcal serotype are determined.
Number of Children (2-5 years of age [YoA]):with serotype specific IgG concentrations for all serotypes included in PCV21 | On day 30
  Ab concentrations for each pneumococcal serotype are measured.
Number of Children/adolescents (6-17 YoA):with serotype specific OPA titers for all serotypes included in PCV21 | On day 30
  Serotype specific OPA titers for each pneumococcal serotype are determined.

SECONDARY OUTCOMES:
Number of Children/adolescents (≥ 2 YoA) with serotype specific OPA titers for all serotypes included in PCV 21 | On day 30
  Serotype specific OPA titers for each pneumococcal serotype are determined.
Number of Children/adolescents (≥ 2 YoA): with serotype specific IgG concentrations for all serotypes included in PCV21 | On day 30
  Ab concentrations for each pneumococcal serotype are measured.
Number of participants (all age groups) with serotype specific IgG concentration ≥ 0.35 μg/mL for all serotypes included in PCV21 | On day 30 after last vaccination
  Ab concentrations for each pneumococcal serotype are measured.
Number of infants (7-11 MoA) and toddlers(12-23 MoA):with serotype specific OPA titers for all serotypes included in PCV21 | On day 30 after last vaccination
  Serotype specific OPA titers for each pneumococcal serotype are determined.
Percentage of infants (7-11 MoA) and toddlers(12-23 MoA): with serotype specific OPA titers ≥ LLOQ for all serotypes included in PCV21 | On day 30 after last vaccination
  Serotype specific OPA titers for each pneumococcal serotype included in the PCV21 formulations are determined. The following threshold values will be considered: ≥ lower limit of quantitation (LLOQ)
Number of Children/adolescents (6-17 YoA):with serotype specific IgG concentrations for all serotypes included in PCV21 | On day 30
  Ab concentrations for each pneumococcal serotype are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations Study Director, Study Director — Sanofi
Locations (38):
- United States (17):
  - Site # 8400008, Paramount, California
  - Site # 8400024, Doral, Florida
  - Site # 8400007, Hialeah, Florida
  - Site # 8400014, Melbourne, Florida
  - Site # 8400009, Miami, Florida
  - Site # 8400016, Miami, Florida
  - Site # 8400021, Fayetteville, Georgia
  - Site # 8400004, Union City, Georgia
  - Site # 8400003, Sioux City, Iowa
  - Site # 8400023, Erlanger, Kentucky
  - Site # 8400018, Biloxi, Mississippi
  - Site # 8400012, Ridgeland, Mississippi
  - Site # 8400002, Omaha, Nebraska
  - Site #8400010, Binghamton, New York
  - Site # 8400025, Rochester, New York
  - Site # 8400001, Houston, Texas
  - Site # 8400017, Stephenville, Texas
- Estonia (7):
  - Site # 2330006, Tallinn, Harju
  - Site # 2330007, Tallinn, Harju
  - Site # 2330002, Tallinn, Harju
  - Site # 2330003, Tallinn, Harju
  - Site # 2330001, Paide, Järvamaa
  - Site # 2330005, Tartu, Tartu
  - Site # 2330004, Tartu
- Poland (7):
  - Site # 6160009, Lodz, Lodskie
  - Site # 6160007, Warsaw, Masovian Voivodeship
  - Site # 6160003, Częstochowa, Silesian Voivodeship
  - Site # 6160002, Bydgoszcz
  - Site # 6160004, Bydgoszcz
  - Site # 6160006, Kłodzko
  - Site # 6160001, Torun
- Thailand (7):
  - Site # 7640002, Hat Yai, Changwat Songkhla
  - Site # 7640003, Mueang Nonthaburi, Chiang Mai
  - Site # 7640008, Bangkok
  - Site # 7640006, Bangkok
  - Site # 7640007, Bangkok
  - Site # 7640004, Chiang Mai
  - Site # 7640001, Pathum Thani

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26551&tenant=MT_SNY_9011